CLINICAL TRIAL: NCT03255317
Title: Developing a Flexible App Data Collection Tool for Substance Use Research
Brief Title: SARA - Substance Abuse Research Assistant
Acronym: SARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Maureen A Walton, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00121553
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Substance Use
Keywords: Substance use, youth, mobile health, data collection adherence, user engagement
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: At each time point at which a participant is eligible to receive an engagement strategy, the participant is randomized to either receive the strategy or not receive the strategy. Participants are only eligible to potentially receive some engagement strategies after completing their self-report survey questions and/or active tasks that day (see "intervention" section for more information).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-participant micro-randomization (Experimental): Intervention includes Reinforcers and Notifications through the app. At each available decision time, each participant is randomly assigned to either receive an engagement strategy or to not receive an engagement strategy.
  Interventions: Behavioral: Reinforcers; Behavioral: Notifications

INTERVENTIONS:
Behavioral: Reinforcers — Memes/Gifs: Immediately after completing their daily ecological momentary assessment using the app, each participant is randomized to receive an inspirational or funny meme or gif that is displayed within the app. Life Insights: Immediately after completing both daily active tasks using the app, each participant is randomized to unlock a life insight. Life insights track data provided by the participant, are stored in a virtual library within the app, and are regularly updated with recent data points.
Behavioral: Notifications — Reminder Push Notifications: All participants receive a push notification reminder from the app at 6pm (the time at which data collection opens) to complete their daily data collection activities. Each day, each participant will be randomized to receive either a generic reminder or a reminder that contains more detailed information (e.g., about upcoming incentives). Inspirational Push Notifications: Each day, each participant will be randomized to receive a push notification at 4pm that contains inspirational song lyrics or celebrity quotes.

SUMMARY:
The aim of this study is to evaluate the efficacy of engagement strategies for increasing daily data collection adherence among substance-using youth between the ages of 14 and 24. The primary hypotheses of this study are that: (1) receiving a reinforcer after completing daily data collection activities will predict next-day completion of targeted data collection activities; and (2) receiving a notification prior to 6pm (when data collection activities open) will predict same-day completion of data collection activities.

DETAILED DESCRIPTION:
Substance use among adolescents and emerging adults remains an alarming public health issue which is associated with the leading causes of death. Although mobile applications are a promising data collection tool for understanding substance use among youth, existing mobile applications are limited in that they are not readily modifiable nor designed for long-term use. To address these challenges, our research team has developed a prototype mobile application named SARA (Substance Abuse Research Assistant) that contains multiple data collection tools (e.g., ecological momentary assessments, active tasks) and features various engagement strategies (reinforcers or notifications) designed to encourage data collection adherence over an extended period of time.

Baseline reinforcers which are administered to all participants include: (1) a virtual aquarium that participants see after opening the app; (2) virtual fish to populate the aquarium, which participants can earn points to unlock by completing daily data collection activities; (3) a new aquarium interface (i.e., leveling up) that participants unlock after using the app for a predetermined amount of time; (4) small financial rewards for each 3-day streak of completing daily data collection activities; and (5) reminder text messages/phone calls from research staff following predetermined reminder schedules. Key reinforcers and notifications are described in detail in the "intervention" section.

This study examines the impact of these key engagement strategies on participant compliance with daily data collection activities over a 30 day field testing period. The primary analyses will use a log linear generalization. The primary longitudinal binary outcome for the reinforcers will be whether on the following day the participant completes one or more self-report validated survey items. The secondary longitudinal binary outcome for the reinforcers will be whether on the following day the participant completes both active tasks. Survey questions answered prior to the randomization as well as the completion of one or more survey questions on the day prior to randomization, and the completion of both active tasks on the day prior to randomization, may be used as control variables in the above analyses of reinforcers. The primary longitudinal binary outcome for the notifications will be whether on the same day the participant completes one or more self-report survey questions. The secondary longitudinal binary outcome for the notifications will be whether on the same day the participant completes both active tasks. The completion of one or more survey questions on the day prior to, and the completion of both active tasks on the day prior to, the randomization will be included as control variables for the notifications.

ELIGIBILITY:
Inclusion criteria:

1. Between the ages of 14 and 24,
2. Has an Android or iPhone smartphone,
3. Self-reported past-month binge drinking (4 drinks for females/5 drinks for males on one occasion) and/or any past-month cannabis use in the absence of a medical marijuana card

Exclusion criteria:

1. Unable to understand English,
2. Not medically stable at intake,
3. Unable to provide informed consent/assent (e.g., cognitively impaired, intoxicated) at intake,
4. Parental consent cannot be obtained at intake (for participants age 14-17),
5. Unable to download the SARA app on smartphone at intake

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Completion of daily self-report survey questions | Same day (2-8 hours later, depending on time of survey completion) for notifications; Next day (24 hours later) for reinforcers.
  Completion of daily self-report survey questions will be measured as "completed' or "not completed." Survey questions include validated items that assess daily mood and substance use. Completed = 1 or more questions answered; not completed = 0 questions answered.

SECONDARY OUTCOMES:
Completion of daily active tasks | Same day (2-8 hours later, depending on time of survey completion) for notifications; Next day (24 hours later) for reinforcers.
  Completion of daily active tasks will be measured as "completed' or "not completed". Completed = 2 tasks; not completed = 1 or 0 tasks

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, MPH, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao P, Klasnja P, Tewari A, Murphy SA. Sample size calculations for micro-randomized trials in mHealth. Stat Med. 2016 May 30;35(12):1944-71. doi: 10.1002/sim.6847. Epub 2015 Dec 28. PMID 26707831
- [Background] Klasnja P, Hekler EB, Shiffman S, Boruvka A, Almirall D, Tewari A, Murphy SA. Microrandomized trials: An experimental design for developing just-in-time adaptive interventions. Health Psychol. 2015 Dec;34S(0):1220-8. doi: 10.1037/hea0000305. PMID 26651463
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Rabbi M, Philyaw-Kotov M, Lee J, Mansour A, Dent L, Wang X, Cunningham R, Bonar E, Nahum-Shani I, Klasnja P, Walton M, Murphy S. SARA: A Mobile App to Engage Users in Health Data Collection. Proc ACM Int Conf Ubiquitous Comput. 2017 Sep;2017:781-789. doi: 10.1145/3123024.3125611. PMID 29503985
- [Derived] Nahum-Shani I, Rabbi M, Yap J, Philyaw-Kotov ML, Klasnja P, Bonar EE, Cunningham RM, Murphy SA, Walton MA. Translating strategies for promoting engagement in mobile health: A proof-of-concept microrandomized trial. Health Psychol. 2021 Dec;40(12):974-987. doi: 10.1037/hea0001101. Epub 2021 Nov 4. PMID 34735165
- [Derived] Rabbi M, Philyaw Kotov M, Cunningham R, Bonar EE, Nahum-Shani I, Klasnja P, Walton M, Murphy S. Toward Increasing Engagement in Substance Use Data Collection: Development of the Substance Abuse Research Assistant App and Protocol for a Microrandomized Trial Using Adolescents and Emerging Adults. JMIR Res Protoc. 2018 Jul 18;7(7):e166. doi: 10.2196/resprot.9850. PMID 30021714